CLINICAL TRIAL: NCT00246363
Title: A Pilot Randomized Placebo-Controlled Trial Designed to Determine the Tolerability and Efficacy of Silymarin (Milk Thistle) vs. Placebo for the Treatment of Chronic Hepatitis C in HIV Infected Patients
Brief Title: A Clinical Research Study Designed To Determine If Treatment of Hepatitis C With Milk Thistle is More Effective Than No Treatment In Patients Infected With Both HIV And Hepatitis C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henry Sacks (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Henry Sacks, MD, PhD, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 02-1185; R21NR008860 (NIH)
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: HIV Infections; Hepatitis C
Keywords: HIV; Hepatitis C
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silymarin (Experimental): Silymarin
  Interventions: Drug: Silymarin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silymarin — Silymarin (milk thistle)
  Arms: Silymarin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
There is some information available that indicates that Milk Thistle is an effective treatment for liver disease. This study will compare Milk Thistle with a placebo, (a medicine that looks just like Milk Thistle but does not contain any Milk Thistle) to see if people with both Hepatitis C and HIV infections show improvement or cure of Hepatitis C. The study will last one year.

DETAILED DESCRIPTION:
Patients with many different diseases are requesting information from health care providers, (physicians and nurses) about alternative therapies. The paucity of evidence based information requires that rigidly structured clinical trials comparing dietary supplements, herbal products and other alternative modalities with either placebo or standard of care be conducted in a timely fashion. There is a body of evidence that Silymarin is both well tolerated and efficacious for the treatment of Hepatitis C. In patients co-infected with HIV & HCV, treatment choices are sometimes limited by intolerable toxicities of standard therapies for the treatment of HCV when combined with antiretroviral therapy for treatment of HIV. This study will seek to determine if Silymarin, an herbal product that is widely used, will be well tolerated and effective in slowing progression of liver damage in patients co-infected with HIV & HCV.

The Informed Consent Document contains all the required elements of informed consent as required by 21CFR50. The consent clearly states that this is research, participation is voluntary and that treatment with Silymarin may not be effective. Every effort has been made to outline whatever is known about any side effects. There are very few. All study participants are followed closely, are given their test results which are also shared with primary care providers. The investigators have convened a Data and Safety Monitoring Board and the Mount Sinai IRB has approved and will monitor the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years old and older
* Blood tests that are positive for a certain type of Hepatitis C known as
* HIV +
* Blood tests for liver function that indicate that the liver is working - must be obtained within one month of study entry
* CD4 counts and HIV viral loads obtained within one month of study entry
* (CD4 count <100 - eligible if HIV Viral Load <25,000)
* (CD4 >100 - eligible with any HIV Viral Load)

Exclusion Criteria:

* Women who are pregnant & breast-feeding & male partners of pregnant women
* Diagnosis of advanced liver disease
* Chronic liver disease other than Hepatitis C
* HIV related infection within two weeks of study entry
* Having had any organ transplant in the past including bone marrow
* History of mental illness including depression within three months of study entry and attempted suicide or hospitalization for the treatment of mental illness at any time in the past
* Chemotherapy treatment or treatment with steroids or other drugs that affect the immune system within six months of study entry
* Problems with alcohol of illegal drugs within one year of study entry. Patients on methadone will be allowed to enter the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
progression of liver damage | one year after enrollment
  progression of liver damage

CONTACTS AND LOCATIONS:
Overall Officials: Henry Sacks, Ph.D., MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.nlm.nih.gov/medlineplus